CLINICAL TRIAL: NCT06740162
Title: A Stage 1 Pilot Test for Feasibility and Efficacy of a Multi-Level Intervention to Increase Physical Activity in Adults With Intellectual Disability: Physical Activity and Community EmPOWERment (PACE)
Brief Title: Physical Activity and Community EmPOWERment Project
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0921; 5R01AG076678-02 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Intellectual Disability; Neurodevelopmental Disorders; Autism Spectrum Disorder; Down Syndrome; Fragile X Syndrome; Cri-du-Chat Syndrome; De Lange Syndrome; Mental Retardation, X-Linked; Prader-Willi Syndrome; Rubinstein-Taybi Syndrome; Trisomy 13 Syndrome; WAGR Syndrome; Williams Syndrome
Keywords: physical activity; intellectual disability; age-associated memory impairment; aging; Alzheimer Disease prevention
MeSH Terms: conditions — Intellectual Disability; Neurodevelopmental Disorders; Autism Spectrum Disorder; Down Syndrome; Fragile X Syndrome; Cri-du-Chat Syndrome; De Lange Syndrome; X-Linked Intellectual Disability; Prader-Willi Syndrome; Rubinstein-Taybi Syndrome; Trisomy 13 Syndrome; WAGR Syndrome; Williams Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE Program (Experimental): The 16-week intervention includes: (1) a weekly group fitness class for adults with ID, (2) web-based training and resources for coaches and exercise professionals; (3) weekly coaching meetings for coaches and adults with ID, and (4) daily/weekly interactions with the PACE interactive web-based dashboard for adults with ID.
  Interventions: Behavioral: PACE Program
- Waitlist Control (No Intervention): Participants assigned to the Waitlist Control Group will not receive any intervention during this interval. Participants will receive the PACE Program after the completion of the 16-weeks for the Intervention Group.

INTERVENTIONS:
Behavioral: PACE Program — The PACE program is a 16-week inclusive exercise program taught and adapted by certified Inclusive Fitness Specialists. Study participants, called athletes, will engage in the fitness class with non-study participants with and without disabilities. Athlete participants will also meet weekly with their coaches (also study participants) to discuss goal setting and interact with the web-based dashboard.
  Arms: PACE Program

SUMMARY:
Purpose: Conduct a wait-list randomized controlled trial (RCT) of an inclusive physical activity program called PACE for adults with intellectual disability (ID) who are not yet showing signs of Alzheimer's Disease (AD)/age-related dementias (ARD).

Participants: Participants include 120 adults with ID, their caregivers, and their coaches (up to 360 individual participants, grouped as triads), recruited through the University of North Carolina at Chapel Hill and the University of Arkansas. Participants also include 16 exercise professionals.

Procedures (methods): Each cohort will include 20 triads who are randomly assigned to the PACE program or the waitlist control group.

DETAILED DESCRIPTION:
Each potential adult with ID or family who contacts the research team will be called and screened for eligibility in the study. To determine eligibility, screening questions will include asking if the adult participant has a formal diagnosis of ID; report of intellectual ability level will be confirmed with direct cognitive testing during the screening assessment visit using scales completed by the participant and caregiver. Also at the screening visit, caregivers will complete the dementia screener for the participants, and participants will be provided with an Actigraph GT9X Link device so they can complete a weeklong physical activity baseline measure. At the second study visit, participants and caregivers will complete the pre-assessments (described below and attached), and participants will have their body composition measured. Questions to all scorable assessments will be required to prevent missing data. Select demographic information will have an additional "prefer not to answer" choice. Participants will complete demographic measures, primary and secondary outcome measures, and feasibility and acceptability measures across the first two study visits. Those who qualify will be randomly assigned to one of two conditions: (1) initial intervention or (2) waitlist control. Individuals assigned to the waitlist control group will begin the intervention after the initial group completes post-assessments.

The 16-week intervention includes: (1) a weekly group fitness class for adults with ID, (2) web based training and resources for coaches and exercise professionals; (3) weekly coaching meetings for coaches and adults with ID, and (4) daily/weekly interactions with the PACE interactive web based dashboard for adults with ID.

A post-assessment visit will be conducted to repeat the pre-assessment measures, and a subset of participants and coaches will also complete an interview to answer open-ended questions about their program experiences. A 12-month follow-up visit will also be scheduled to measure body composition again.

Brief description of measures to be completed by Caregivers as follows:

Vineland Adaptive Behavior Scales-3: (VABS) (Vineland-3) is a standardized assessment tool that utilizes semi-structured interview to measure adaptive behavior and support the diagnosis of intellectual and developmental disabilities, autism, and developmental delays. Interviews are expected to take 1-2 hours and will take place during the screening visit.

National Task Group-Early Detection Screen for Dementia: (NTG-EDSD) This measure was adapted from the Dementia Screening Questionnaire for Individuals with Intellectual Disabilities (DSQIID) and can be used for the early detection screening of those adults with an intellectual disability who are suspected of or may be showing early signs of mild cognitive impairment or dementia. The NTG-EDSD is not an assessment or diagnostic instrument, but an administrative screen that can be used by staff and family caregivers to note functional decline and health problems and record information useful for further assessment. This assessment will take place during the screening visit.

Add Health Wave 5 Questionnaire: Questions will be used from the Wave 5 Survey including questions on background (biological sex, gender, race/ethnicity), health and health care (co-occurring conditions and medical treatments, illness and physical limitations, and fitness tracking (experiences using fitness tracking devices, current exercise habits). This measure will take place during the pre and post study visits.

Waisman Activities of Daily Living (W-ADL): The W-ADL is a caregiver-report that measures activities of daily living and assesses functioning. It has demonstrated high internal consistency (Cronbach alphas= .88-.94) and reliability over time (Kappas= .92-.93) in adults with ID. This measure will take place during the pre and post study visits.

Brief description of adult with ID measures as follows:

The Leiter-3: is a widely used nonverbal measure of intelligence and cognitive abilities that is suitable to use for individuals with cognitive delays, speech or hearing problems, Attention Deficit Hyperactivity Disorder (ADHD), or traumatic brain injury. The battery subtest scores are converted to a scaled score and the sum of the scaled scores yields a nonverbal intelligence quotient (IQ)/composite score. This assessment will take place during the screening visit.

World Health Organization Quality of Life Brief Version Assessment (WHOQoL-BREF and WHO Disabilities Module): The WHOQoL-BREF and WHO Disabilities module is an abbreviated 39-item version of the original WHOQOL tool that has been used in adults with ID. The domain scores will be used to measure the general quality of life (Overall, Health, Physical, Psychological, Social, Environment, and Disabilities Module). This measure will take place during the pre and post study visits.

NIH-Toolbox Cognitive Battery (NIHTB-CB): The NIHTB-CB will measure mental and cognitive functioning. It has been validated in individuals with ID and adults across the spectrum of Alzheimer's disease and age-related cognitive decline. It is an iPad-based assessment of memory, executive function, and crystallized intelligence. This measure will take place during the pre and post study visits.

NIH-Toolbox Emotional Battery: The NIHTB-EB will measure emotional health across several domains: Psychological Well-Being, Social Relationships, Stress and Self-Efficacy, and Negative Affect. This is an iPad-based assessment that will take place during the pre and post study visits.

Physical Activity Measures: These measures will take place during the pre and post study visits.

Grip strength (NIH Toolbox): This test consists of squeezing the hand dynamometer for a 1-rep max strength assessment.

The 4-Stage Balance Test: This test consists of four standing positions that are progressively harder to maintain.

30-Second Chair Stand: This test consists of participants getting up from a chair without using their arms. They get up and sit down repeatedly for 30 seconds. Their score is the number of times they can get up from the chair

Timed Up & Go (TUG): This test consists of participants getting up from a chair, walking 10 feet across the room around a cone, and sitting back down.

2-Minute Walk Endurance: This test consists of participants walking as fast as they can for two-minutes up and down the hallway of the assessment spaces.

Bod Pod: This scan will measure body composition using Air Displacement Plethysmograph (ADP). Participants at the University of North Carolina site will be briefed on the Bod Pod and sit inside for up to 5 minutes. This measure will take place during the pre- and post-study visits, as well as the one-year follow-up visit.

DXA Scan: This scan will measure body composition using dual energy X-ray absorptiometry. Participants at the University of Arkansas site will be briefed and lay on the DXA scan table for around 15 minutes. This measure will take place during the pre- and post-study visits, as well as the one-year follow-up visit. Participants who are pregnant, think they may be pregnant, or have had unprotected sex in the last 30 days will not receive a DXA scan.

ELIGIBILITY:
Inclusion criteria for adults with ID will include:

* ages 18 and older with a prior clinical diagnosis of ID, confirmed by scores < 70 and + 90% on the Leiter-3 International Performance Scales and/or an adaptive behavior measure using the Vineland Adaptive Behavior Scales,
* Medical clearance to participate in moderate-to-vigorous physical activity as determined by the American College of Sports Medicine (ACSM) preparticipation algorithm,
* Adult does not show clinically elevated symptoms of Alzheimer's Disease (AD)/ Alzheimer's Disease and Related Dementias (ADRD) as indicated by a score of < 20 on the Dementia Screening Questionnaire for Individuals with Intellectual Disabilities.
* One caregiver/guardian is able and willing to participate.
* must tolerate at least 8 hours of daily wear-time of Actigraph device during initial assessment period (4 of 7 days),
* must average 20 minutes or less of moderate to vigorous physical activity (MVPA) minutes per day (140 MVPA minutes or less across 7-day period measured during the initial assessment period, and
* must reside in North Carolina or Arkansas.

Exclusion Criteria for adults with ID:

• Diagnosis of AD, dementia, or related disorders. Participants will not be excluded based on gender, race, or ethnicity. There will be no upper age limit due to the heterogeneity of onset of AD/ADRD in individuals with ID.

Inclusion criteria for coach will include:

* access to the internet and a mobile device,
* has weekly contact with the adult participant with ID,
* can converse and read in English to comprehend intervention materials and website content, and
* must reside in North Carolina or Arkansas

Inclusion criteria for caregiver will include:

* ability to converse and read in English to comprehend and answer interview questions, (2) must care for an adult with ID who is willing to participate in the study,
* must reside in North Carolina or Arkansas, and
* must attend all study visits with adult with ID.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Steps Per Day as Measured by the ActiGraph GT9X Link | Baseline, post-intervention (16 weeks)
  The Actigraph GT9X Links measures daily step counts. Step counts less than 2500 are classified as basal, step counts between 2500 to 4999 are classified as limited, step counts between 5000 to 7499 are classified as low, step counts between 7500-9999 are classified as somewhat active, step counts between 10000 to 12499 are classified as active, and step counts over 12500 are classified as very active.
Minutes of Moderate-to-Vigorous Activity Per Day as Measured by the ActiGraph GT9X Link | Baseline, post-intervention (16 weeks)
  The Actigraph GT9X Links measures activity counts each minute of wear time. Each activity count over 3,941 equals 1 minute of moderate-vigorous physical activity. A total of 150 or more weekly MVPA minutes meets Physical Activity guideline recommendations.

SECONDARY OUTCOMES:
Body Composition from Baseline as Measured by percentage of total body mass | Baseline, post-intervention (16 weeks), Follow-up (74 weeks)
  Body composition will be assessed using the Bod Pod at University of North Carolina and the DXA at University of Arkansas. The Bod Pod is an air displacement plethysmograph that uses whole-body densitometry to determine fat, lean, and total body mass. Total body mass >30%for men/40% for women=risky, 21- 30%for men/31-40%for women=extra fat, 13-20%for men/23-30% for women=acceptable, 9-12% for men/19 -22% for women=excellent health ), 5-8 % for men/15-18 %for women= ultra lean, and <5 percent and <15%=risky low body fat. The Dual-Energy X-Ray Absorptiometry (DXA) scan measures body fat percentage. Optimal body fat percentages for adults age 20-29 are 16-24%for females/7-17 % for males; age 30-39 are 17-25% for females/12-21% for males, age 40-49 are 19-28% for females/14-23% for males, ages 50-59 are 22-31% for females/16-24% for males, age 60+ are 22-33% for females/17-25% for males. Numbers that are higher than optimal=overweight and lower than optimal=underweight.
Wellbeing from Baseline as Measured by the World Health Organization Quality of Life Assessment and Disabilities Module | Baseline, post-intervention (16 weeks)
  Adults with intellectual disability (ID) will complete the World Health Organization Quality of Life Assessment and World Health Organization Disabilities Module measures of quality of life. The WHOQoL-BREF and WHO Disabilities module is an abbreviated 39-item version of the original WHOQOL tool that has been used in adults with ID. The domain scores will be used to measure the general quality of life (Overall, Health, Physical, Psychological, Social, Environment, and Disabilities Module). Scores Range from 0-100 with higher scores indicating better quality of life.
Daily Living Skills from Baseline as Measured by the Waisman Activities of Daily Living Scale | Baseline, post-intervention (16 weeks)
  Activities of daily living will be measured using caregiver-report using the Waisman Activities of Daily Living (W-ADL). The 17-item W-ADL measures the level of independence in performing typical daily activities for adolescents and adults. The W-ADL has demonstrated high internal consistency (Cronbach alphas= .88-.94) and reliability over time (Kappas= .92-.93) in adults with intellectual disability. Performance is rated on a 3-point scale (0 means the participant does not do the activity at all, 1 means the participant does the activity with help, and 2 means the participant does the activity independently). The scoring range is 0 to 34 with higher scores signifying greater independence in daily living activities.
Mental and Cognitive Functioning from Baseline as Measured by the NIH-Toolbox Cognitive Battery | Baseline, post-intervention (16 weeks)
  Mental and cognitive functioning will be measured using the NIH-Toolbox Cognitive Battery (NIHTB-CB), which has been validated in individuals with intellectual disability and adults across the spectrum of Alzheimer's disease and age-related cognitive decline. The NIHTB-CB is an iPad-based assessment of memory, executive function, and crystallized intelligence. The Fluid Cognition Composite includes fluid ability measures: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. The Crystallized Cognition Composite Score includes the Picture Vocabulary and Reading Tests. The composite scores are derived by averaging the standard scores of each of the measures. Higher scores indicate higher levels of functioning - a score at/near 100 indicates ability that is average compared with others nationally, 115 suggests above-average, 130 suggests superior ability, 85 suggests significantly below-average, and a score of below suggests very low.
Psychological Well-Being, and Social Relationships from Baseline as Measured by the NIH Toolbox Emotion Battery | Baseline, post-intervention (16 weeks)
  Social belonging will be assessed through questionnaires using the NIH Toolbox Emotion battery including the Psychological Well-Being, Social Relationships domains with adults with intellectual disability. The NIH-Toolbox Emotion Battery has been validated in adults with and without neurological disorders. The Psychological Well-Being Domain is derived from a weighted average of T-scores for Positive Affect, General Life Satisfaction, and Meaning & Purpose. Higher scores indicate more self-reported psychological well-being. Scores below 40 suggest low levels of psychological well-being, and scores above 60 suggest high levels of psychological well-being. The Social Satisfaction summary score is derived from Friendship, Loneliness, Emotional Support, Instrumental Support, and Perceived Rejection. Higher scores indicate higher social satisfaction. Scores below 40 suggest low levels of social satisfaction, and scores above 60 suggest high levels of social satisfaction.
Stress and Self-Efficacy, and Negative Affect from Baseline as Measured by the NIH Toolbox Emotion Battery | Baseline, post-intervention (16 weeks)
  Social belonging will be assessed through questionnaires using the NIH Toolbox Emotion battery including the Stress and Self-Efficacy, and Negative Affect domains. Stress and Self-Efficacy focus on individual perceptions about the nature of their events and their relationship to the perceived coping resources. On Perceived Stress, higher scores are indicative of more perceived stress. Scores at or below 40 suggest low perceived stress and scores at or above 60 suggest high perceived stress. On Self-efficacy, higher scores are indicative of more general self-efficacy. Scores at or below 40 suggest low self-efficacy levels and scores at or above 60 suggest high self-efficacy levels. Negative Affect summary score is derived from the Anger-Affect, Anger-Hostility, Sadness, Fear-Affect, and Perceived Stress Domains. Higher scores are indicative of more negative affect. Scores at or below 40 suggest low levels, and scores at or above 60 suggest high levels of negative affect.
Grip Strength from Baseline as Measured by the Hand Dynamometer | Baseline, post-intervention (16 weeks)
  Grip strength will be assessed by a 1-rep max strength assessment. Participants will be asked to squeeze the hand dynamometer as hard as they can for 3 seconds. Grip strength is measured with a standard score metric (normative mean = 100, Standard Deviation = 15). It compares the performance of the test-taker to those in the entire NIH Toolbox nationally representative normative sample. Higher standard scores indicate better performance.
Ability to Maintain Balance from Baseline as Measured by the 4-Stage Balance Test | Baseline, post-intervention (16 weeks)
  Balance will be measured by the 4-Stage Balance Test. The test consists of four standing positions that are progressively harder to maintain. Each position is held for a maximum of 10 seconds. This is scored by number of seconds, with 10 being the maximum score indicating static balance.
Functional Lower Extremity Strength and Endurance from Baseline as Measured by the 30-Second Chair Stand | Baseline, post-intervention (16 weeks)
  Functional strength will be measured by the 30-second chair stand. This test consists of participants getting up from a chair without using their arms. They get up and sit down repeatedly for 30 seconds. Their score is the number of times they can get up from the chair. The higher the score indicates greater leg strength and endurance.
Mobility from Baseline as Measured by the Timed Up & Go (TUG) | Baseline, post-intervention (16 weeks)
  Mobility will be assessed through the Timed Up & Go (TUG) assessment. This test consists of participants getting up from a chair, walking 10 feet across the room around a cone, and sitting back down. This is scored in seconds. A time of ≥12 seconds to complete the TUG is at risk for falling.
Endurance from Baseline as Measured by the 2-Minute Walk Endurance Test | Baseline, post-intervention (16 weeks)
  This test consists of participants walking as fast as they can for two-minutes up and down the hallway of the assessment spaces. The participant's raw score is the distance walked in two minutes, reported in feet (and fractions thereof). This score is then converted to the NIH Toolbox normative scores. Higher scores are indicative of better endurance. Scores at or below 30 are suggestive of motor dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Brianne R Tomaszewski, PhD., MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of Arkansas, Fayetteville, Arkansas
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Savage MN, Tomaszewski BT, Hume KA. Step It Up: Increasing Physical Activity for Adults With Autism Spectrum Disorder and Intellectual Disability Using Supported Self-Management and Fitbit Technology. Focus Autism Other Dev Disabl. Published online January 25, 2022:108835762110737. doi:10.1177/10883576211073700
- [Background] Diaz KM. Leisure-time physical activity and all-cause mortality among adults with intellectual disability: the National Health Interview Survey. J Intellect Disabil Res. 2020 Feb;64(2):180-184. doi: 10.1111/jir.12695. Epub 2019 Dec 2. PMID 31788881
- [Background] De la Rosa A, Olaso-Gonzalez G, Arc-Chagnaud C, Millan F, Salvador-Pascual A, Garcia-Lucerga C, Blasco-Lafarga C, Garcia-Dominguez E, Carretero A, Correas AG, Vina J, Gomez-Cabrera MC. Physical exercise in the prevention and treatment of Alzheimer's disease. J Sport Health Sci. 2020 Sep;9(5):394-404. doi: 10.1016/j.jshs.2020.01.004. Epub 2020 Feb 4. PMID 32780691
- [Background] Sinai A, Bohnen I, Strydom A. Older adults with intellectual disability. Curr Opin Psychiatry. 2012 Sep;25(5):359-64. doi: 10.1097/YCO.0b013e328355ab26. PMID 22744404
- [Background] Shooshtari S, Martens PJ, Burchill CA, Dik N, Naghipur S. Prevalence of Depression and Dementia among Adults with Developmental Disabilities in Manitoba, Canada. Int J Family Med. 2011;2011:319574. doi: 10.1155/2011/319574. Epub 2011 Aug 8. PMID 22295184
- [Background] McCallion P, McCarron M. Ageing and intellectual disabilities: a review of recent literature. Curr Opin Psychiatry. 2004;17(5):349-352. doi:10.1097/01.yco.0000139968.14695.95
- See also: Study recruitment and participant interaction website — https://mypaceprogram.org/